CLINICAL TRIAL: NCT00680641
Title: The Effects of Simvastatin in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Simvastatin in Chronic Obstructive Pulmonary Disease (COPD)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of East Anglia (Other)
Responsible Party: Dr Andrew M Wilson, University of East Anglia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2007RESP06
Record Dates: First submitted 2008-05-16; First posted 2008-05-20 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2011-08

CONDITIONS: COPD; Emphysema
Keywords: COPD; Emphysema; Simvastatin
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Simvastatin 40mg
  Interventions: Drug: Simvastatin
- B (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Simvastatin — 40mg of Simvastatin once daily
  Arms: A
Drug: Placebo — 40mg of placebo once daily
  Arms: B

SUMMARY:
To determine the effects of 2 months therapy with simvastatin 40mg once per day compared to placebo in a double-blind placebo-controlled study of patients with COPD.

DETAILED DESCRIPTION:
Statins (HMG-Coenzyme A reductase inhibitors) are widely used clinically as lipid lowering drugs; however they have also been shown to exhibit anti-inflammatory and anti-oxidant properties(1). Recently published large retrospective cohort studies, in patients with chronic obstructive pulmonary disease (COPD), suggest that statins reduce mortality and COPD related admissions(2). Possible mechanisms of action include effects on cell adhesion molecules, changes in inflammatory mediator release, antioxidant effect and increased clearance of apoptoic cells. Simvastatin has been shown to reduce the development of smoking induced emphysema in rats with reductions in MMP-9 activity and simvastatin withdrawal leads to increased MMP levels in hypercholesterolaemic patients. Serum concentrations of TNFa and high sensitive C Reactive protein(3) (hs-CRP) are reduced with simvastatin therapy in patients with hypercholesterolaemia and risk of cardiovascular disease respectively. No clinical trial has directly evaluated the clinical effects of statins in patients with COPD in terms of induced sputum MMP profile, alveolar nitric oxide or pulmonary physiology.

We have modified our published method of RNA purification, developed to purify RNA from cartilage, tendon or synovium(4), to yield good quality RNA from sputum with relative simplicity and low cost. We have identified MMP-2, -9 and -14 in the sputum of healthy volunteers (unpublished pilot data) and will utilise this technique in the current study. Exhaled breath condensate (EBC) is completely non-invasive, requires no co-operation from individuals and provides information about a number of inflammatory and oxidation pathways. Markers of oxidative stress (8-isoprostane and hydrogen peroxide) and nitric oxide products can be measured in exhale breath condensate(5) and are related to disease activity in patients with COPD. Markers of oxidative stress increase in concentration in EBC during exacerbations of COPD are reduced after treatment with the antioxidant N-acetyl cysteine(6). Hydrogen peroxide is not stable and therefore 8-isoprostane is a preferable marker of oxidative stress unless the sample is measured on line.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged more than 45 years.
* Physician labelled diagnosis of chronic obstructive pulmonary disease,emphysema or chronic bronchitis.
* Smoker or ex-smoker with a pack year smoking history of greater than 20 pack years
* FEV1 30-70% predicted
* FEV1/FVC< 70%
* Body Mass Index <25kg/m2

Exclusion Criteria:

* 1. Cardiac or pulmonary disease other than chronic obstructive pulmonary disease.
* Untreated hypothyroidism
* Respiratory infection defined as fever, nasal/sinus congestion, fatigue, cough, antibiotic use or yellow/green sputum within 4 weeks prior to study.
* Receiving current oral corticosteroid therapy or leukotriene modifying therapy.
* Severe or uncontrolled co-morbid disease
* History of atopy or asthma
* Clinical history of bronchiectasis
* Pregnancy or breastfeeding
* Women of child-bearing potential, unless adequate contraception is used (ie contraceptive pill or double-barrier contraception - partner using condom and subject using spermicide, diaphragm, intra-uterine device or contraceptive sponge)
* Unable to give written informed consent
* Patients receiving a statin prior to entry into the study
* Hypersensitivity to simvastatin or to any of the excipients.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-04; Primary Completion 2011-02 (Actual); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
The difference in serum high sensitivity C-reactive protein (HsCRP) between simvastatin and placebo | 4 checks over a four month period at 2 weeks, 10 weeks, 14 weeks and 22 weeks.

SECONDARY OUTCOMES:
The difference between treatment with simvastatin and placebo for Clinical COPD Questionnaire | 4 months
The difference between treatment with simvastatin and placebo for Spirometry - FEV1, FVC, FEV1/FVC ratio | 4 months
The difference between treatment with simvastatin and placebo for Induced sputum differential cell count | 4 months
The difference between treatment with simvastatin and placebo for Induced sputum mRNA for MMP and TIMPs | 4 months
The difference between treatment with simvastatin and placebo for Exhaled breath condensate 8-isoprostane concentration | 4 Months
The difference between treatment with simvastatin and placebo for Serum TNFa | 4 months
The difference between treatment with simvastatin and placebo for Cholesterol | 4 Months

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Wilson, MD, MRCP (UK), Principal Investigator — Clinical Senior Lecturer, University of East Anglia
Locations (2):
- United Kingdom (2):
  - CRTU University of East Anglia, Norwich, Norfolk
  - CRTU Norfolk and Norwich University Hospital, Norwich, Norfolk

REFERENCES:
- [Background] Hothersall E, McSharry C, Thomson NC. Potential therapeutic role for statins in respiratory disease. Thorax. 2006 Aug;61(8):729-34. doi: 10.1136/thx.2005.057976. PMID 16877692
- [Background] Soyseth V, Brekke PH, Smith P, Omland T. Statin use is associated with reduced mortality in COPD. Eur Respir J. 2007 Feb;29(2):279-83. doi: 10.1183/09031936.00106406. Epub 2006 Oct 18. PMID 17050558
- [Background] Hanefeld M, Marx N, Pfutzner A, Baurecht W, Lubben G, Karagiannis E, Stier U, Forst T. Anti-inflammatory effects of pioglitazone and/or simvastatin in high cardiovascular risk patients with elevated high sensitivity C-reactive protein: the PIOSTAT Study. J Am Coll Cardiol. 2007 Jan 23;49(3):290-7. doi: 10.1016/j.jacc.2006.08.054. Epub 2007 Jan 8. PMID 17239709
- [Background] Kevorkian L, Young DA, Darrah C, Donell ST, Shepstone L, Porter S, Brockbank SM, Edwards DR, Parker AE, Clark IM. Expression profiling of metalloproteinases and their inhibitors in cartilage. Arthritis Rheum. 2004 Jan;50(1):131-41. doi: 10.1002/art.11433. PMID 14730609
- [Background] Montuschi P. Exhaled breath condensate analysis in patients with COPD. Clin Chim Acta. 2005 Jun;356(1-2):22-34. doi: 10.1016/j.cccn.2005.01.012. Epub 2005 Mar 23. PMID 15936301
- [Background] Kasielski M, Nowak D. Long-term administration of N-acetylcysteine decreases hydrogen peroxide exhalation in subjects with chronic obstructive pulmonary disease. Respir Med. 2001 Jun;95(6):448-56. doi: 10.1053/rmed.2001.1066. PMID 11421501
- [Background] van der Molen T, Willemse BW, Schokker S, ten Hacken NH, Postma DS, Juniper EF. Development, validity and responsiveness of the Clinical COPD Questionnaire. Health Qual Life Outcomes. 2003 Apr 28;1:13. doi: 10.1186/1477-7525-1-13. PMID 12773199
- [Background] Pizzichini E, Pizzichini MM, Efthimiadis A, Evans S, Morris MM, Squillace D, Gleich GJ, Dolovich J, Hargreave FE. Indices of airway inflammation in induced sputum: reproducibility and validity of cell and fluid-phase measurements. Am J Respir Crit Care Med. 1996 Aug;154(2 Pt 1):308-17. doi: 10.1164/ajrccm.154.2.8756799.
- [Background] Standardization of spirometry--1987 update. Statement of the American Thoracic Society. Am Rev Respir Dis. 1987 Nov;136(5):1285-98. doi: 10.1164/ajrccm/136.5.1285. No abstract available. PMID 3674589